CLINICAL TRIAL: NCT05903508
Title: Comparative Effect of Functional Task Training Versus Function Therapy Program on Gross Motor Function, Range of Motion and Balance in Children With Cerebral Palsy
Brief Title: Comparative Effect of Functional Task Training Versus Function Therapy Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0703
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy
Keywords: gross motor function, cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Its a randomized control trial,used to evaluate the comparative affect of functional task training versus functional therapy programsm on gross motor function, range of motion on, and balance in cerebral palsy children.Subject with hemiplagic Cerebral palsy (GMFCS level 1-11) meeting the predetermined inclusion and exclusion criteria will be divided into two groups using simple random sampling technique
Who Masked: Participant
Masking Description: Participant will get seperate treatment protocol and possible efforts will be put to mask the both groups about thier treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional task training Group. (Active Comparator): In this group patients will performed functional task training program was performed including non-walking (i-iii) and walking activities: (i) standing from a seated position; (ii) reaching for an object overhead, which required ankle plantar flexion from the standing position, and returning to the initial position with the heel leaning on the floor; (iii) stepping on and off a bench; (iv) walking up and down stairs; and (v) walking on flat surfaces and ramps. for 8 weeks, 50 minutes per day, 3 times per week. The individual session lasted approximately 10 minutes including the rest intervals.
  Interventions: Other: Functional task training and functional therapy program; Other: Functional therapy program Group
- functional therapy program (Active Comparator): In this group patients will performed functional therapy program as goal directed training to optimize the child to practice goal including stand when turning around between chair, cycles 5m on stationary bicyle on smooth surface, kicking a ball during 8 weeks, the children practiced a goal in 50 mintute per day and 3 times a week.
  Interventions: Other: Functional task training and functional therapy program; Other: Functional therapy program Group

INTERVENTIONS:
Other: Functional task training and functional therapy program — Functional task training group this will receive walking and no walking activities
Other: Functional therapy program Group — Functional therapy program Group this will receive goal directed training

SUMMARY:
cerebral palsy is the brain injury or brain malformation occur before, during and immediately after birth (while brain is still under development) and its effect muscle tone, reflexes, posture coordination gross and fine motor skill and oral motor functioning. The functional training is the physiotherapist and occupational therapy rehabilitation technique focus on strength and function of musculoskeletal system and its help the patients to making their daily life activity easier. The functional task training program consisted of non-walking (i-iii) and walking (iv-v) activities: (i) standing from a seated position; (ii) reaching for an object overhead, which required ankle plantar flexion from the standing position, and returning to the initial position with the heel leaning on the floor; (iii) stepping on and off a bench; (iv) walking up and down stairs; and (v) walking on flat surfaces and ramps. Children with cerebral palsy frequently receive. functional therapy programs the children participated in activities pertaining to everyday skills such as eating, playing, communication, and mobility. To optimize the child's opportunities to practice towards the goals, parents and preschool staff were guided on efficiently encouraging the child. Support and instructions from the professional to help them to develop better motor skills and increase independence in tasks like self-care, play, and recreational activities.so the study aimsto improve balance, gross motor function, and range of motion by using these functional training task and functional therapy program. In my study compare the compare task training versus functional therapy programsm on gross motor function, range of motion on, and balance in cerebral palsy children.

DETAILED DESCRIPTION:
The randomized control trial will be conducted through convenient sampling. There will be two group the experimental group will receive functional task training. according to GMFS, Pediatric balance scale and goniometer to assess the gross motor function, ROM and balance in cerebral palsy, while control group will receive functional therapy program (bobath technique) to improve gross motor function, ROM and balance in cerebral palsy. The duration of the treatment will be 8 weeks. Gross motor function, pediatric balance scale, and goniometer will be used as outcome measure. Data will be analyzed on spss version 29, normality of the data will be checked and test will be applied according to the normality of the data either in will be parametric test or nonparametric based on the normality

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* GMFCS (Gross Motor Function Classification System) score is in between 1-2,
* Ability to follow command
* Cerebral palsy diagnosed child (
* Age 6-12yr

Exclusion Criteria:

* • Deformity like scoliosis. pelvic, oblique, and hip deformity

  * Age more than 16
  * Visual disorder
  * Mental retardation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Goniomete | 8 weeks
  It will measure range of motion
Pediatric balance scale | 8 weeks
  it is 14 items that measure the balance in the context of everyday task in pediatric population in 3 domain sitting standing and changing of position
Gross Motor Function Measure scale | 8 weeks
  . The GMFM-88 item scores can be summed to calculate raw and percent scores for each of the five GMFM dimensions of interest selected goal areas and total GMFM-88 scores. The scoring system of the GMFM is a four-point scale divided into five categories (lying and rolling; sitting; crawling and kneeling; standing; walking, running)

CONTACTS AND LOCATIONS:
Overall Officials: kinza Naeem, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sah AK, Balaji GK, Agrahara S. Effects of Task-oriented Activities Based on Neurodevelopmental Therapy Principles on Trunk Control, Balance, and Gross Motor Function in Children with Spastic Diplegic Cerebral Palsy: A Single-blinded Randomized Clinical Trial. J Pediatr Neurosci. 2019 Jul-Sep;14(3):120-126. doi: 10.4103/jpn.JPN_35_19. Epub 2019 Sep 27. PMID 31649770